CLINICAL TRIAL: NCT06567262
Title: Oral Health Related Quality of Life and Cost Effectiveness in CAD/CAM and Conventional Metallic Partial Denture Frameworks in Mandibular Kennedy Class III Cases: A Randomised Cross-over Trial
Brief Title: Compare CAD/CAM Metallic RPD to Conventional Metallic RPD in Terms of Oral Health Related Quality of Life
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Tarek Salah Hashim Ali, assistant lecturer, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5724
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Partial Edentulism Class 3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD/CAM metallic removable partial denture (Experimental): CAD/CAM technology will be used to scan the oral cavity to create a 3D model that can be digitally surveyed. After designing RPD digitally by computer software, wax pattern can be constructed by milling or rapid prototyping technology. This wax pattern would be cast conventionally into RPD framework.
  Interventions: Device: CAD/CAM metallic removable partial denture
- Conventional metallic removable partial denture (Active Comparator): Conventional RPD design involves the production of stone casts, geometric characterization of the tooth and soft tissues related to the path of insertion, and careful designation of RPD components (major and minor connectors, rests, clasps, and base retention) using a direct waxing method.
  Interventions: Device: Conventional metallic removable partial denture

INTERVENTIONS:
Device: CAD/CAM metallic removable partial denture — Make digital scans using an intraoral scanning device. Scan the maxillary (antagonistic scan) and mandibular (pre-preparation scan) arches, as well as an initial digital record of the inter-occlusal relation (occlusal scan).
  Analyse the digital cast using CAD software. Primary electronic surveying will be carried out to ensure if the tooth preparations will be needed.
  Make a definitive intraoral scan only of the prepared teeth and record the maxillary-mandibular relationship.
  The virtual cast is digitally surveyed and the design of the framework is done using computer software. The wax pattern 3D framework information will be converted into a standard tessellation language (STL) file and transfer to a rapid prototyping (RP) system to be printed and finally cast using the conventional technique to produce RPD framework.
  Arms: CAD/CAM metallic removable partial denture
Device: Conventional metallic removable partial denture — Primary impressions will be taken, the impressions will be poured to construct a study casts.
  Maxillary Face-bow record and diagnostic bite will be taken. The study casts will be mounted on semi adjustable articulator to check inter-arch space.
  Surveying of the study cast will be done. Required mouth preparation will be carried out then secondary impression will be taken using special tray.
  Secondary impression will be poured to obtain master cast which will be surveyed to confirm proper mouth preparation, blocked out and then wax pattern will be designed and constructed.
  A metallic framework will be obtained using the conventional lost wax technique and casting.
  Intraoral try in of the framework will be done followed by bite registration record.
  The next step will be teeth setting and try in. Heat cured acrylic resin denture base will be processed, finished and polished conventionally.
  Arms: Conventional metallic removable partial denture

SUMMARY:
Patients will be randomised to receive CAD/CAM metallic removable partial denture (RPD) followed by Conventional metallic RPD (Group A), or the opposite sequence (Group B), with a 3-month wear duration for each denture and washout period for one week. Patients will be recalled at base line and 3 months following prosthetic insertion to evaluate Oral health related quality of life. It is hypothesized that removable partial dentures with CAD/CAM metallic RPD frameworks would improve Oral health related quality of life than those with Conventional metallic RPD frameworks.

DETAILED DESCRIPTION:
Eligible patient will be selected from outpatient clinic in removable prosthodontics department clinic. Patients will be informed of the nature of the research work and informed consent will be obtained from each of them. Only motivated patients who shows cooperation will participate in the study. Patients will be randomised to receive CAD/CAM metallic RPD followed by Conventional metallic RPD (Group A), or the opposite sequence (Group B), with a 3-month wear duration for each denture and washout period for one week. Patients will be recalled at base line and 3 months following prosthetic insertion to evaluate Oral health related quality of life and cost effectiveness.

Patients will be subjected to:

* Comprehensive clinical examination and understanding of patient's chief complaints and their expectations from the prosthesis.
* Digital periapical radiographs with paralleling technique will be taken for the abutment teeth as base line for bone height before prosthesis construction.

CAD/CAM metallic RPD:

1. Make digital scans using an intraoral scanning device. Scan the maxillary (antagonistic scan) and mandibular (pre-preparation scan) arches, as well as an initial digital record of the inter-occlusal relation (occlusal scan).
2. Analyse the digital cast using CAD software. Primary electronic surveying will be carried out to ensure if the tooth preparations will be needed.
3. Make a definitive intraoral scan only of the prepared teeth and record the maxillary-mandibular relationship.
4. The virtual cast is digitally surveyed and the design of the framework is done using computer software. The wax pattern 3D framework information will be converted into a standard tessellation language (STL) file and transfer to a rapid prototyping (RP) system to be printed and finally cast using the conventional technique to produce RPD framework.
5. The overall treatments costs, including the fees from the dental laboratory, will be calculated and compared with the costs of a conventionally fabricated RPD.

Conventional metallic RPD:

1. Primary impressions will be taken using irreversible hydrocolloid impression material (alginate), the impressions will be poured to construct a study casts.
2. Maxillary Face-bow record and diagnostic bite will be taken. The study casts will be mounted on semi adjustable articulator to check inter-arch space.
3. Surveying of the study cast will be done. Required mouth preparation will be carried out then secondary impression will be taken using special tray.
4. Secondary impression will be poured to obtain master cast which will be surveyed to confirm proper mouth preparation, blocked out and then wax pattern will be designed and constructed.
5. A metallic framework will be obtained using the conventional lost wax technique and casting.
6. After de-investing, finishing and polishing, the framework will be fitted on the master cast. Intraoral try in of the framework will be done followed by bite registration record.
7. The next step will be teeth setting and try in. Heat cured acrylic resin denture base will be processed, finished and polished conventionally.
8. The finished removable partial denture will then be checked intraorally for any needed modifications and finally delivered.

Criteria for discontinuing or modifying intervention:

Regardless of any decision to modify their assigned intervention, study participants will be retained in the trial whenever possible to enable follow up data collection and prevent missing data. If periodontitis is reported during follow up period, a suitable mouthwash will be given to the patient, who will be recalled regularly to closely observe the changes. If periodontitis continue, patient will be advised to stop wearing the prosthesis for two weeks till inflammation subsides and supra and sub gingival scaling and root planning will be carried out. Continued bone loss or inflammation might dictate trial discontinuation. If inflammation related to fitting surface of the denture or to any of the components was reported during follow up period, the RPD will be checked for any pressure areas to be relieved, a suitable mouthwash will be given to the patient and as mentioned before; the patient will be recalled regularly to closely observe the changes. The period of discontinuing the treatment will be included in the follow up period.

Strategies to improve adherence to intervention:

The patients will be asked to attend regular follow up visits and their adherence to the oral hygiene instructions will be monitored. Any signs of inflammation as redness or profuse plaque will be photographed and shown to the patient. This will reflect the importance of the oral hygiene measures.

Patients will receive phone calls from secretary to remind him/her of the follow up visits. Address of the patients will be recorded, in case the patient did not show up a home visit will be considered.

Patients will be recalled at one and 3 months after RPD insertion and whenever they have a complaint.

Sample size:

The investigators are planning a study of a continuous response variable from matched pairs of study subjects. Prior data indicate that the difference in the response of matched pairs is normally distributed with a standard deviation of 25.7. If the true difference in the mean response of matched pairs is 15, the investigators will need to study 19 pairs of subjects to be able to reject the null hypothesis that this response difference is zero with probability (power) 0.8. The Type I error probability associated with this test of this null hypothesis is 0.05.

Recruitment:

1. Fresh Patient attending in the outpatient clinic in faculty of dentistry, Cairo University will be enrolled in the study.
2. The department patients' database will be reviewed and possible candidates for the trial will be called.

Another eligibility examination will be made by the researcher and the research will be discussed with all patients and only motivated patient will join the research.

B) Assignment of interventions

Allocation:

1. Randomization:

   * Method of random sequence generation (computerized random number generator).
   * Allocation ratio (1:1)
   * Type of randomization: simple
   * Randomization sequence will be kept with (HF)
2. Allocation concealment mechanism:

   Every participant will grasp an opaque sealed opaque envelop from a box. The envelope will contain a number that corresponds to the treatment. Being opaque and sealed ensures allocation concealment.
3. Implementation (HF) is the person who will generate the allocation sequence centrally and who is responsible for ensuring proper randomization and allocation concealment.

Masking/blinding:

Care provider, participants, and statistician will be blinded.

C) Data collection, management, and analysis:

Data collection methods:

Plans for assessment and collection of outcome:

The collected data whether personal or numerical will be stored on excel sheets as an electronic copy and printed hard copy sheets. The primary outcome data will be collected before RPD insertion as baseline and then after insertion with one month and 3 months. While, the secondary outcome data will be collected before RPD insertion. Treatment will be coded in the questionnaire as A & B.

Plans to promote participant retention and complete follow-up:

* Telephone numbers and address of all subjects in the study will be recorded as a part of the signed consent
* All subjects will receive a phone call at the time of the predetermined follow up dates.
* Paying transportation fees.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unilateral bounded saddles in the mandible (Kennedy class III).
2. Opposing dentition is fully intact or restored.
3. Sufficient inter-arch space.
4. Angle's class I maxilla-mandibular relationship.

Exclusion Criteria:

1. Periodontal affection of the abutment teeth.
2. Skeletal mal-relation.
3. Unmotivated patients to maintain adequate oral hygiene to follow up.
4. Patients with neuromuscular and Psychiatric disorders.
5. Systematic disease affecting bone and periodontal health.
6. Insufficient inter-arch space.
7. Patients with physical reasons that could affect follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Oral health related quality of life | 3 months
  Oral health related quality of life will be measured by a valid and reliable questionnaire which is Oral health impact profile questionnaire (OHIP) before RPD insertion then after RPD insertion with one and 3 months for both groups. It consists of 5 questions representing the four suggested dimensions: Oral Function, Orofacial Pain, Orofacial Appearance and Psychosocial Impact. Questions were made on a 5-point Likert scale (0 = never; 1 = hardly ever; 2 = occasionally; 3 = fairly often; and 4 = very often).

SECONDARY OUTCOMES:
Cost effectiveness | 3 months
  Cost effectiveness analysis - The incremental cost-effectiveness ratio (ICER) will be calculated using the following formula: ICER = direct cost difference / outcome score difference between CAD/CAM metallic RPD and Conventional metallic RPD
  - ICER indicates an additional cost that needs to increase extra one unit in each outcome measure with CAD/CAM metallic RPD comparing to Conventional metallic RPD treatment

IPD SHARING:
Plan to Share IPD: No